CLINICAL TRIAL: NCT00443313
Title: HPV Testing to Improve Cervical Cancer Screening in the Mississippi Delta (Mississippi Delta Project)
Brief Title: Human Papillomavirus (HPV) Testing to Improve Cervical Cancer Screening in the Mississippi Delta
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907080; 07-C-N080
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-06-25

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervical neoplasia; Screening; HPV; Cervical Cancer Screening
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

* Cancer of the cervix (bottom third of the uterus, or womb) can be prevented by regular Pap tests (also called Pap smears), which check for changes in the cells of the cervix. Because many women in the United States have regular Pap smears, cervical cancer is not common in this country. However, the disease is common among women in the Mississippi Delta because of poor participation in screening programs.
* The major causes of cervical cancer are persistent human papillomaviruses (HPV) infection by cancer-associated HPV types and lack of screening. These viruses cause an infection that often goes away by itself, but if it does not go away, over a long time lead to cervical cancer. HPV causes cervical abnormalities, which are detected by Pap smears and then treated.

Objectives:

-To determine whether an at-home self-collection method for obtaining cells from the cervix can be a simple, safe and inexpensive way to screen for cervical cancer for women who don t go to the health clinic regularly.

Eligibility:

* Women who reside in the counties of Leflore, Sunflower, Washington or Tallahatchie, Mississippi.
* Women between 26 and 65 years of age who are not pregnant and who have not had a hysterectomy.

Design:

Screening study participants undergo the following:

* The doctor takes a cervical sample using the same self-collection device that women will use at home to self-collect.
* Pelvic examination and Pap test. For this test, the woman lies on an exam table and the doctor inserts an instrument called a speculum into the vagina, opening it to see the cervix. A special brush is used to take a few cells from the cervix. The cells are placed on a glass slide and sent to a lab for examination.
* Cervical cell specimen collection using an at-home self-collection kit that participants will use at home after 2 weeks
* At-home self-collection by participant after 2 weeks.
* Referral to a doctor for follow-up care, if needed.
* Colposcopy (see below) in all women with a Pap test that is abnormal or positive for HPV and for some women with a normal smear.

Colposcopy study participants undergo the following:

* The doctor takes a cervical sample using the same self-collection device that women will use at home to self-collect.
* Colposcopy, an exam in which the doctor examines the cervix using a light and looks through a magnifying device to see if there is any abnormal tissue on the cervix. During this exam, the doctor may remove a small sample of tissue to diagnose any abnormality. Participants also have a sample collected using the self-collection kit.
* At-home cervical sample collection by participant after 2 weeks.
* Notification if further medical care is required and treatment if the biopsy looks abnormal.

DETAILED DESCRIPTION:
Background: Cytology screening programs have effectively reduced cervical cancer incidence and mortality in the U.S. by greater than 75%. However, these programs requiring repeated clinician-administered Pap smears do not adequately cover medically-underserved populations. Based partly on HREB/DCEG etiologic research, we now know that carcinogenic types of human papillomavirus (HPV) cause virtually all cases of cervical cancer. Supported by our translational work with DCP, HPV DNA testing is already approved by the FDA as an adjunctive screening modality to cytology in this country and as a primary screening modality to cytology in this country and as a primary screening modality internationally. A validated screening program of HPV DNA testing of self-collected cervicovaginal specimens would permit wider coverage screening than cytology in the populations underserved by cytology-based testing like the Mississippi Delta region.

Objective: To assess the technical feasibility (i.e. non-inferiority or equivalence to cytology for detection of cervical precancer and cancer) of cervical cancer screening based on self-collection and HPV DNA testing of cervicovaginal specimens from women aged greater than or equal to 30 years old who live in the Mississippi Delta.

Methods: One thousand women will be enrolled during 18 months, including 500 attending colposcopy due to cytologic abnormality, 250 women who regularly attend a screening clinic, and 250 unscreened women who have not had a Pap smear within the last 3 years (according to current screening guidelines) but recruited to attend a screening. Three clinical specimens will be collected from each woman. A cervicovaginal specimen (for HPV testing) and a cervical specimen (for cytology and HPV testing) will be collected from each woman by the physician. At the time of the clinic visit women will be give a kit for self-collection of a second cervicovaginal specimen (for HPV testing) to be returned by mail within two weeks. All three specimens from each woman will be tested by two clinical DNA tests that use pooled-probes for detection of carcinogenic HPV: an FDA-approved signal amplification test (Hybrid Capture 2 from Digene) and a new DNA amplification test (AMPLICOR from Roche) currently in clinical trials. Specimens will also be tested retrospectively by a research PCR asay that detects 37 HPV types, which will help us evaluate the performance of the two clinical HPV tests. Women attending their screening visit who test positive by cytology (atypical squamous cells of undetermined significance or worse) or for carcinogenic HPV will be referred to colposcopy along with a random sample of HPV negative, cytologic negative women (n equals 100).

Analysis: We will compare the clinical performance of HPV DNA testing of self-collected specimens to that of cytology (at a threshold of atypical squamous cells of unknown significance (ASCUS) or more severe) for detection of histologically confirmed cervical intraepithelial neoplasia grade 2 (CIN2) or more severe (greater than or equal to CIN2). Cytology results will be based on standard-of-care cytology screening for women attending the screening visit and repeat cytology for women attending colposcopy. An estimated 150 cases of greater than or equal to CIN2 will be identified. This is an equivalence study, where we wish to reject the null hypothesis that HPV self-testing is greater than 10% less sensitive than cytology. Assuming cytology has a 75% sensitivity for greater than or equal to CIN2, a sample size of 150 subjects has 84% power (alpha=0.05) (one-sided non-inferiority or equivalence test of correlated proportions) to rule out a 10% decrement in sensitivity for self-collection with HPV DNA testing compared with cytology will guide whether the new technique could be broadly introduced for cervical cancer screening.

ELIGIBILITY:
* INCLUSION CRITERIA:

Five-hundred women attending colposcopy and 500 women receiving cytology screening, including 250 unscreened women, will be recruited for the study. Non-pregnant, non-hysterectomized women aged 26-65 will be recruited.

EXCLUSION CRITERIA:

Women under 26 or over 65 years of age.

Pregnant women or women having given birth to a child in the past 8 weeks. To insure women included in the study are not pregnant, we will ask women during the consenting process if they are pregnant. Women who answer yes for either query will be excluded. Participants will also receive a reminder call for their 2-week self-collection. At that time, women again will be asked if they are pregnant. If any woman answers yes, she will be instructed to not self-collect.

Women who have had a total hysterectomy.

Women who have an overt cancerous lesion visible upon exam by the clinician.

Other reasons to exclude women include the inability to speak English, the appearance of mental incompetence, or refusal to participate or sign the informed consent form.

Ages: 26 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2007-01-24; Study Completion 2015-06-25

PRIMARY OUTCOMES:
Detection CIN II+ | During course of study

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Gage, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Harper DM, Franco EL, Wheeler C, Ferris DG, Jenkins D, Schuind A, Zahaf T, Innis B, Naud P, De Carvalho NS, Roteli-Martins CM, Teixeira J, Blatter MM, Korn AP, Quint W, Dubin G; GlaxoSmithKline HPV Vaccine Study Group. Efficacy of a bivalent L1 virus-like particle vaccine in prevention of infection with human papillomavirus types 16 and 18 in young women: a randomised controlled trial. Lancet. 2004 Nov 13-19;364(9447):1757-65. doi: 10.1016/S0140-6736(04)17398-4. PMID 15541448
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Smigal C, Thun MJ. Cancer statistics, 2006. CA Cancer J Clin. 2006 Mar-Apr;56(2):106-30. doi: 10.3322/canjclin.56.2.106. PMID 16514137
- [Background] Wang SS, Sherman ME, Hildesheim A, Lacey JV Jr, Devesa S. Cervical adenocarcinoma and squamous cell carcinoma incidence trends among white women and black women in the United States for 1976-2000. Cancer. 2004 Mar 1;100(5):1035-44. doi: 10.1002/cncr.20064. PMID 14983500